CLINICAL TRIAL: NCT02577926
Title: Ruxolitinib Versus Best Available Therapy in Patients With High-risk Polycythemia Vera or High-risk Essential Thrombocythemia - The Ruxo-BEAT Trial
Brief Title: The Ruxo-BEAT Trial in Patients With High-risk Polycythemia Vera or High-risk Essential Thrombocythemia
Acronym: Ruxo-BEAT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-181
Record Dates: First submitted 2015-10-01; First posted 2015-10-16 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Polycythemia Vera (PV); Essential Thrombocythemia (ET)
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential | interventions — ruxolitinib; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Ruxolitinib (Experimental): Ruxolitinib will be administered orally at a dose of 10 mg twice daily (both PV and ET) for two consecutive years.
  Interventions: Drug: Ruxolitinib
- Best available therapy (BAT) (Active Comparator): BAT may include all currently used treatment options. BAT is at the choice of the investigator (monotherapy with i.e. hydroxyurea, anagrelide, interferon, busulfan, immunomodulators etc). BAT will be administrated for two consecutive years.
  Interventions: Drug: BAT

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is a JAK1/2-specific tyrosine kinase inhibitor (TKI) which has been approved for the treatment of symptomatic myelofibrosis. The compound was shown to be superior to hydroxyurea in reducing splenomegaly and constitutional symptoms.
  Other Names: Study drug; Jakavi
  Arms: Ruxolitinib
Drug: BAT — BAT is at the choice of the investigator (monotherapy with i.e. hydroxyurea, anagrelide, interferon, busulfan, immunomodulators etc).
  Other Names: Control Treatment
  Arms: Best available therapy (BAT)

SUMMARY:
The Philadelphia chromosome negative myeloproliferative neoplasms (MPN) comprise a group of clonal hematological malignancies that are characterized by chronic myeloproliferation, splenomegaly, different degrees of bone marrow fibrosis, and disease-related symptoms including pruritus, night sweats, fever, weight loss, cachexia, and diarrhea. In addition, due to elevated numbers of leucocytes, erythrocytes and/or platelets, the disease course can be complicated by thromboembolic disease, hemorrhage, and leukemic transformation as well as myelofibrosis.

Patients with polycythemia vera (PV) typically harbor an increased number of blood cells from all three hematopoietic cell lineages due to clonal amplification of hematopoetic stem cells, while patients with essential thrombocythemia (ET) typically show a predominant expansion of the megakaryocytic lineage. Most patients with PV below the age of 60 years are currently being treated with acetylsalicylic acid +/- phlebotomy only, and patients with low-risk ET have an almost normal life expectancy and often do not require specific treatment. However, PV- as well as ET-patients with a higher risk for complications require cytoreductive treatment. In addition, constitutional symptoms can be unbearable to patients even in the absence of bona fide high risk factors, and these patients may similarly benefit from antineoplastic therapy.

DETAILED DESCRIPTION:
Polycythemia vera (PV) and essential thrombocythemia (ET) are classical Philadelphia-negative myeloproliferative neoplasms (MPN) that are characterized by an excess of cells in the peripheral blood, clonal bone marrow hyperplasia, and extramedullary hematopoiesis. The symptoms of these patients may range from asymptomatic disease to symptomatic disease that may significantly affect their activities of daily living, such as severe generalized pruritus, night sweats and fevers, erythromelalgia, bone and muscle pain, weight loss, and fatigue. Moreover, the patients may develop thromboembolic and hemorrhagic complications, transition to myelofibrosis (MF), and transformation to acute leukemia. In principle, the only potentially curative therapy for MPNs is allogenic stem cell transplantation (allo-SCT). However, due to significant transplant-associated morbidity and mortality, this therapeutic option is only applied in exceptional cases of ET or PV. The majority of patients do not qualify for allo-SCT since the risks of this treatment clearly outweigh the potential benefits. Moreover, even with a non-transplantation approach, patients with ET and PV have a life expectancy comparable to or close to healthy age-matched control persons. For patients with standard risk PV, phlebotomy and acetylsalicylic acid are standard of care (target hematocrit below 45 %), while patients with standard risk ET should receive either no specific treatment or acetylsalicylic acid (provided that no microvascular symptoms or secondary acquired von Willebrand syndrome are present).

However, in patients who are at high risk to develop thromboembolic or hemorrhagic complications (high-risk patients), cytoreductive treatment is generally indicated to prevent these potentially life-threatening complications. In PV and ET, high risk patients are characterized by advanced age (> 60 years) and / or a history of thromboembolic or hemorrhagic events {1,2,3}. In ET, a platelet count > 1500 x 109/l is associated with an increased risk of bleeding, and thus should result in a platelet lowering treatment {2}. In PV, in addition to the risk-score based therapy, cytoreduction is also required in patients with progressive or marked myeloproliferation (leukocytosis, thrombocytosis, symptomatic splenomegaly, increase of frequency of phlebotomy requirement), or devastating constitutional symptoms {1,2,4}. In Germany, best available therapy (BAT) includes approved drugs such as hydroxyurea (HU; approved for both PV and ET) and anagrelide (approved for second-line treatment of ET) and non-approved options such as alpha-interferon, pipobroman, busulfan (in elderly patients), and radioactive phosphorus (32P). In rare cases, patients may also benefit from splenic irradiation or splenectomy.

Ruxolitinib is a JAK1/2-specific tyrosine kinase inhibitor (TKI) which has been approved for the treatment of symptomatic myelofibrosis. The compound was shown to be superior to hydroxyurea in reducing splenomegaly and constitutional symptoms. Ruxolitinib is currently studied in phase 2 and phase 3 clinical trials for HU-resistant or HU-intolerant PV and ET. The aim of the present study is to assess the feasibility, efficacy, and safety of ruxolitinib treatment vs. BAT in patients with high-risk PV or -ET.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to studyspecific procedures or assessments which are not routinely performed for diagnosis or monitoring of PV or ET, and the subjects must be willing to comply with treatment and to follow up assessments and procedures
2. Patient must be 18 years of age or older
3. Patient´s ECOG performance status must be 0-2
4. Patient must fulfill WHO 2008 diagnostic criteria for either polycythemia vera (PV) or essential thrombocythemia (ET). Moreover, PV- and ET-patients have to be classified as high risk according to defined criteria.

   For patients with high risk PV OR PV with indication for cytoreductive therapy due to progressive myeloproliferation, AT LEAST ONE of the following must be fulfilled (according to DGHO onkopedia) (Barbui, et al., 2011). (Passamonti, 2009):
   * Age > 60 years
   * Previous documented thrombosis or thromboembolism
   * Platelet count > 1500 x 109/L
   * Poor tolerance of phlebotomy or frequent phlebotomy requirement
   * Symptomatic or progressive splenomegaly
   * Severe disease-related symptoms (according to the investigators definition)
   * Progressive leukocytosis with leukocyte count > 20 x 109/L

   For patients with high risk ET, AT LEAST ONE of the following must be fulfilled (according to DGHO guidelines):
   * Age > 60 years
   * Platelet count> 1500 x 109/L
   * Previous thrombosis or thromboembolism
   * Previous severe hemorrhage related to ET (defined as decrease of Hgb of at least 2 g/dl)
5. Patients must fulfill the following criteria regarding prior therapy:

   PV patients:

   Never treated with cytoreductive drugs except hydroyurea, anagrelide, or interferon for up to 6 weeks maximum (phlebotomy and/or aspirin are allowed)

   ET patients:

   Naïve and pretreated patients may be entered in this trial.
6. Patient must have adequate liver function as indicated by a total bilirubin, AST, and ALT ≤ 2 of the institutional upper limit of normal (ULN) value, unless directly attributable to the patient's MPN
7. Patient must have a creatinine clearance >40ml/min calculated according to the modified formula of Cockcroft and Gault, eGFR, or directly measured after 24h-urine collection
8. Patients must be able to swallow and retain oral medication

Exclusion Criteria:

1. Patients who meet criteria for post PV-MF or post ET-MF (IWG-MRT)
2. Patients who have received previous ruxolitinib treatment
3. Patients who have a history of anaphylaxis following exposure to the BAT drug of choice
4. Patients who have an inadequate bone marrow reserve as demonstrated by ANC ≤ 1 x 109/l OR platelet count <50 x 109/l
5. Patients who have known hepatitis B or C or HIV infection
6. Patients who suffer from other severe, concurrent diseases, including tuberculosis, serious cardiac functional dysfunction (class III or IV as defined by the New York Heart Association Classification), uncontrolled diabetes, uncontrolled hypertension, severe pulmonary disease (i.e. COPD with hypoxemia), or major organ malfunction that could interfere with the patient's ability to participate in the study
7. Patients who have history of active substance or alcohol abuse within the last year
8. Female patients who are pregnant or nursing
9. Patients who have participated in another interventional trial and/or used investigational agents or concurrent anticancer treatment for concomitant disease within the last 4 weeks of registration
10. Any circumstance at the time of study entry that would preclude completion of the study or the required follow-up prohibits inclusion into this study
11. Subjects who have had an active malignancy during the previous 3 years except for treated cervical intraepithelial neoplasia, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin, each with no evidence for recurrence in the past 3 years
12. Patients who have uncontrolled bacterial, viral, or fungal infection
13. Patients who have any medical condition requiring prolonged use of oral corticosteroids with a dose of more than 20 mg per day (> 1 month)
14. Patients who have severe cerebral dysfunction and/or legal incapacity
15. Patients who have had active splanchnic vein thrombosis within the last 3 months (includes Budd-Chiari, portal vein, splenic and mesenteric thrombosis)
16. Patients who have thyroid dysfunction which is not adequately controlled
17. Fertile men or women of childbearing potential cannot be included unless they are:

    * surgically sterile or > 2 years after the onset of menopause and/or
    * willing to use a highly effective contraceptive method (Pearl Index <1) such as oral contraceptives, intrauterine device, sexual abstinence, or barrier method of contraception (i.e. condoms) in conjunction with spermicidal jelly during study treatment
18. Patients who are taking any of the following prohibited medication:

    * clarithromycin, telithromycin, troleandomycin (antibiotics)
    * ritonavir, indinavir, saquinavir, nelfinavir, amprenavir, lopinavir (HIV protease inhibitors)
    * itraconazole, ketoconazole, voriconazole, fluconazole (antifungals)
19. Patients with a diagnosis of galactose or lactose intolerance or a glucose-galactose- malabsortion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The rate of complete clinicohematologic response rate (CHR) as defined by Barosi et al 2009 | at month 6

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | at month 6 and 12
The complete response rate (CR) at month 6 as defined by Barosi et al Blood 2013 (revised ELN response criteria) | month 6
The rate of complete responses (CHR) at month 12 as defined by Barosi et al Blood 2009 | month 12
The efficacy as assessed by the absence of phlebotomy (Hct <45%) | through study completion, an average of 2 years
The efficacy as assessed by the reduction in spleen size (palpable spleen that is reduced by > 50% from baseline measured by palpation and ultrasound) OR platelet count < 600 x 10^9/l (ET) | through study completion, an average of 2 years
Proportion of subjects achieving both durable absence of phlebotomy eligibility AND durable spleen volume reduction measured by palpation and ultrasound (PV) OR durable platelet count <600 x 10^9/l (ET) (durable defined as >3 months) {Barosi et al 2013) | through study completion, an average of 2 years
The rate of overall clinicohematologic remissions (CR + PR) according to both guidelines (Barosi et al 2009 and 2013) | through study completion, an average of 2 years
Safety of both regimen | through study completion, an average of 2 years
  Adverse events will be assessed according to CTCAE 4.0 throughout the study until 30 days after EoT for patients in both regimens

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Koschmieder, Prof. Dr., Principal Investigator — RWTH University Hospital MK4
Locations (23):
- Germany (23):
  - Universitätsmedizin Mannheim III. Medizinische Klinik Hämatologie und Internistische Onkologie, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Ulm Klinik für Innere Medizin III, Ulm, Baden-Wurttemberg
  - Rems-Murr Klinikum Winnenden, Winnenden, Baden-Wurttemberg
  - Studienzentrum Aschaffenburg, Aschaffenburg, Bavaria
  - III. Medizinischen Klinik des Klinikums rechts der Isar der TU München, Müchen, Bavaria
  - Klinikum Nürnberg Nord Medizinische Klinik 5, Nuremberg, Bavaria
  - Universitätsklinikum Hamburg Eppendorf Klinik und Poliklinik für Onkologie, Hämatologie und KMT mit Sektion Pneumologie, Hamburg, Hamburg
  - Universitätsmedizin Mainz III. Medizinische Klinik und Poliklinik, Mainz, Hesse
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Bonn Medizinische Klinik und Poliklinik III, Bonn, North Rhine-Westphalia
  - Johanniter-Krankenhaus Rheinhausen GmbH Hämatologie / Internistische Onkologie / Tagesklinik, Duisburg, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf Klinik für Hämatologie, Onkologie und Klinische Immunologie, Düsseldorf, North Rhine-Westphalia
  - Marienhospital, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen Klinik für Hämatologie, Essen, North Rhine-Westphalia
  - Mühlenkreiskliniken Johannes Wesling Klinikum Minden Klinik für Hämatologie, Onkologie und Palliativmedizin, Minden, North Rhine-Westphalia
  - Universitätsklinikum Magdeburg, Magdeburg, Sachesen-Anhalt
  - Klinikum Chemnitz gGmbH Klinik für Innere Medizin III, Chemnitz, Saxony
  - Universitätsklinikum Dresden Medizinische Klinik und Poliklinik I, Dresden, Saxony
  - Universitätsklinikum Halle (Saale), Halle, Saxony-Anhalt
  - Charite Universitätsmedizin Berlin; Medizinische Klinik m.S. Hämatologie, Onkologie und Tumorimmunologie, Berlin
  - Universitätsklinikum Freiburg - Klinik für Innere Medizin I, Freiburg im Breisgau
  - Universitätsklinik Jena - Klinik für Innere Medizin II, Jena
  - UNIVERSITÄTSKLINIKUM Schleswig-Holstein - Klinik für Hämatologie und Onkologie, Campus Lübeck, Lübeck

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isfort S, Manz K, Teichmann LL, Crysandt M, Burchert A, Hochhaus A, Saussele S, Kiani A, Gothert JR, Illmer T, Schafhausen P, Al-Ali HK, Stegelmann F, Hanel M, Pfeiffer T, Giagounidis A, Franke GN, Koschmieder S, Fabarius A, Ernst T, Warnken-Uhlich M, Wolber U, Kohn D, Pfirrmann M, Wolf D, Brummendorf TH; German CML study group. Step-in dosing of bosutinib in pts with chronic phase chronic myeloid leukemia (CML) after second-generation tyrosine kinase inhibitor (TKI) therapy: results of the Bosutinib Dose Optimization (BODO) Study. Ann Hematol. 2023 Oct;102(10):2741-2752. doi: 10.1007/s00277-023-05394-0. Epub 2023 Aug 18. PMID 37592092
- [Derived] Koschmieder S, Isfort S, Wolf D, Heidel FH, Hochhaus A, Schafhausen P, Griesshammer M, Wolleschak D, Platzbecker U, Dohner K, Jost PJ, Parmentier S, Schaich M, von Bubnoff N, Stegelmann F, Maurer A, Crysandt M, Gezer D, Kortmann M, Franklin J, Frank J, Hellmich M, Brummendorf TH; German Study Group for Myeloproliferative Neoplasms (GSG-MPN). Efficacy and safety of ruxolitinib in patients with newly-diagnosed polycythemia vera: futility analysis of the RuxoBEAT clinical trial of the GSG-MPN study group. Ann Hematol. 2023 Feb;102(2):349-358. doi: 10.1007/s00277-022-05080-7. Epub 2022 Dec 23. PMID 36564535